CLINICAL TRIAL: NCT02344979
Title: The Study of rHuTPO/rHuIL-11 in the Treatment for Chemotherapy-induced Thrombocytopenia in Patients With NSCLC Receiving Gemcitabine and Cisplatin or Carboplatin Chemotherapy
Brief Title: The Study of rHuTPO/rHuIL-11 in the Treatment for Chemotherapy-induced Thrombocytopenia in Patients With NSCLC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: ShenyangSunshine
Record Dates: First submitted 2015-01-18; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Thrombocytopenia
Keywords: NSCLC; Chemotherapy; thrombocytopenia; rhTPO
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Randomized, open label, controlled, parallel, multi-center Study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group rHuTPO: Patients were treated with recombinant human thrombopoietin(rHuTPO)on d2,d4,d6,d9 of chemotherapy cycle.
- Group rHuIL-11: Patients were treated with recombinant human interleukin-11(rHuIL-11)on d9-d15 after chemotherapy.

SUMMARY:
Purpose: To evaluate the efficacy and safety of rHuTPO/rHuIL-11 in the treatment for chemotherapy-induced thrombocytopenia in patients with NSCLC receiving gemcitabine and cisplatin or carboplatin chemotherapy.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Patients aged 18 years -75 years, male or female;
2. histologically or cytologically confirmed non-small cell lung cancer;
3. consistent with the indication of chemotherapy
4. the decrease of platelets appeared in the screen chemotherapy period and the platelet count is less than 50 * 109/ L;
5. the expected survival was more than 3 months;
6. patients must have the ability to understand and the willingness to sign a written informed consent;
7. to be able to follow the study and follow-up procedures

Exclusion Criteria:

1. pregnant or lactating women;
2. patients who had severe allergic history on biological preparation;
3. the existing serious acute infection without control;
4. Patients receiving radiotherapy;
5. more than 3 metastatic tumor of bone were found in the screening period, and the platelet count did not restore to 100 * 109/ L on the screening period on the seventeenth day of the screening period;
6. with a history of pulmonary embolism, myocardial infarction patients, thrombus history of thrombosis or activity in the past 3 months;
7. Sepsis, disseminated intravascular coagulation (DIC); hypersplenism or any other illness sickness that can exacerbate thrombocytopenia appeared in the previous cycles of chemotherapy;
8. tumor metastasis was found in the central nervous system;

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years, Male or females
* Patients with NSCLC for whom treatment with gemcitabine and cisplatin or carboplatin
* Platele counts ≤ 50×109/L during Screening chemo cycle
* ECOG PS score is ≤ 2
* The predicted life expectancy ≥3 months
* Written informed consent

Exclusion Criteria:

* Pregnant or nursing women
* Known history of severe anaphylactic reaction to biologics
* Uncontrolled severe infection
* History of bone or central nervous system metastasis
* History of platelet disorder
* Active bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC for whom treatment with gemcitabine and cisplatin or carboplatin,and Platele counts ≤ 50×109/L during Screening chemo cycle
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
The mean minimal and maximal platelet count after rHuTPO or rHuIL-11. | 28days

SECONDARY OUTCOMES:
The time to achieve platelet count ≥75×109/L and ≥100×109/L after rHuTPO or rHuIL-11. The duration of platelet count <50×109/L after rHuTPO or rHuIL-11. | 28days
The number of platelet transfusions after rHuTPO or rHuIL-11. | 28days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- See also: Related Info — http://www.3sbio.com